CLINICAL TRIAL: NCT06222957
Title: The Effects of HER2 Receptor Signaling on Human Brown Fat Activity: A 1-year Prospective Cohort Study in Trastuzumab-treated Breast Cancer Patients Versus HER2 Negative Controls
Brief Title: The Effects of HER2 Receptor Signaling on Human Brown Fat Activity
Acronym: HEAT
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Tora Ida Henriksen, Primary Investigator, Rigshospitalet, Denmark
Other Study IDs: H-23055495
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: HER2 receptor; HER2 receptor positive; Brown adipose tissue; Human brown fat; Trastuzumab; Cooling; Infrared thermography
MeSH Terms: conditions — Breast Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will draw blood samples, but not for genetic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HER2 positive group: HER2-positive (HER2+) and Estrogen receptor-positive (ER+) breast cancer patients undergoing adjuvant chemotherapy including trastuzumab.
  Interventions: Other: None (Observational study)
- Control group: HER2-negative breast cancer patients (HER2-) and Estrogen receptor-positive (ER+) breast cancer patients undergoing adjuvant chemotherapy without trastuzumab.
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — Both groups recieve standard care as decided by the responsible clinicians at the department of Oncology. The course of the treatment is completely independent from the observations in the present study.

SUMMARY:
The objective of this observational study is to investigate the significance of the HER2 receptor for brown fat activity in humans. Our preliminary data clearly demonstrates that the ErbB signaling pathway, which includes the HER2 receptor, strongly promotes development and function of cultured human BAT cells. The HER2 receptor is a part of the ErbB signaling pathway, and antibodies against thee HER2 receptor are a part of the standard treatment for HER2-positive breast cancer. Therefore, the hypothesis is that the activity of brown fat will be reduced in patients treated with HER2 blocking antibody compared to patients who are not treated with HER2 blocking antibody. The present study simply takes advantage of the treatment protocol to explore the contribution of the HER2 receptor in the development of brown adipose tissue in humans. Participants will complete two testing days, one before and one after their treatment period of approx. one year. On the testing days, identification of brown fat activity will be performed using cooling and infrared thermography. In addition, resting metabolic rate and a glucose tolerance test will be performed. Since presence of active brown adipose tissue in humans is inversely related to obesity, total and visceral fat mass, plasma glucose levels, presence of cardiovascular disease and diabetes status, it is of great importance to investigate the molecular mechanisms for development of brown fat tissue and may lead to discovery of novel strategies to counteract obesity and obesity related disorders.

DETAILED DESCRIPTION:
BACKGROUND:

Breast cancer is the most common cancer among women worldwide, and with increasing survival rates focus on long-term adverse effects of treatment has increased. Weight gain is well documented and common occurrence for many breast cancer patients. Recently, a review reported that 50-96% of women experience weight gain during treatment. Furthermore, many patients report a progressive weight gain in the months and years after treatment and patients rarely return to their pre-diagnosis weight. Moreover, weight gain in breast cancer patients has been linked to a poor prognosis compared to patients without weight gain, and to obesity-related disorders including metabolic syndrome.

Adipose tissue is one of the largest human organs. Two functionally distinct types of adipose tissue exist: white adipose tissue and brown adipose tissue (BAT). While BAT was long thought to be present only in rodents and human infants, it is now clear that active BAT also exists in varying degrees in adult humans. Activated BAT has great capacity for energy consumption and takes up large amounts of blood lipids and glucose to use in thermogenesis, and the presence of active BAT in humans is inversely related to obesity, total and visceral fat mass, plasma glucose levels, presence of cardiovascular disease and diabetes status. In accordance, acute cooling increases energy expenditure compared to thermoneutral conditions and correlates with higher BAT activity. Finding ways to activate BAT in humans is thus an attractive approach to prevent weight gain and ensuing comorbidities.

Human epidermal growth factor receptor 2 (HER2) positive breast cancer accounts for ~15 % of breast cancer cases, and direct inhibition of the HER2 receptor (also called the ErbB2 receptor) is used as standard treatment of HER2-positive breast cancer.

Our preliminary data clearly demonstrates that the ErbB signaling pathway, which includes the HER2 receptor, strongly promotes development and function of cultured human BAT cells and mouse brown adipose tissue. A potential secondary effect of the HER2 receptor blockade used in cancer treatment, is the binding of these inhibitors to ErbB2 receptors in the adipose tissue subsequently affecting downstream signaling pathways that might influence the activity of brown adipose tissue and thereby whole-body metabolism. In support of this hypothesis, weight gain during chemotherapy in HER2-positive breast cancer patients is associated with a decrease in the activity of brown adipose tissue.

Since BAT activity has been suggested as a target to limit weight gain and metabolic disorders, it is of great importance to understand the molecular mechanisms behind BAT recruitment and function in humans. This study will provide insight into the contribution of the HER2 receptor in the development of brown adipose tissue in humans and may thus lead to discovery of novel strategies to counteract obesity and obesity related disorders in breast cancer survivors as well as in the general population.

STUDY SET-UP

Against this background, a prospective cohort study will be performed at the Centre for Physical Activity (CFAS), and the Department of Oncology, both located at Rigshospitalet, Copenhagen, Denmark. A total of 30 patients will be recruited. This includes patients with breast cancer HER2+/ Estrogen receptor (ER)+ treated with the recombinant monoclonal anti-neoplastic antibody combination trastuzumab (n = 15) and BMI and age-matched HER2-/ER+ patients with breast cancer, who are not treated with ErbB2/HER2 receptor blockage, will be used as a control group (n = 15). The treatment is planned and initiated according to standard of care and for clinical reasons. The present study simply takes advantage of the treatment protocol to explore a physiological mechanism, hence participation in the study does not affect the treatment regimen. After cessation of the study period subjects will continue their treatment as prescribed by the oncologists prior to study enrolment.

Patients included in the study will undergo two identical test days; one prior to the treatment and one by the end of the treatment. The study does not include any additional interventions, restrictions, or investigations during the treatment period. For each testing day, the participants will be assessed for body composition (DXA scan) and anthropometrics. This will be followed by a cooling protocol to activate the brown adipose tissue. BAT activity will be measured by infrared thermography. Furthermore, participants will undergo measurements of resting metabolic rate, an oral glucose tolerance (OGTT) test and blood samples.

Provided that the patient fulfilled the inclusion criterion concerning cold activated BAT (see inclusion criteria), they will be invited to a second test day after adjuvant treatment. This test day will be similar to the first, i.e., including anthropometric measurements, a DXA scan, blood samples, an OGTT, indirect calorimetry measurements, a cooling intervention and IRT assessment of BAT activity.

AIM

The objective of this project is thus to investigate the effects of HER2 blockade on human brown adipose tissue activity in HER2+ breast cancer patients as well as associated metabolic parameters.

Secondarily, the study aim to investigate whether a decrease in BAT activity is associated with weight gain or increased fat mass (as assessed by DXA-scan), decreased metabolic rate and changes in metabolic parameters including glycemic control in patients treated with HER2 blocking antibodies.

HYPOTHESIS

The hypothesis is that the activity of brown fat will be reduced in patients treated with HER2 blocking antibody trastuzumab for 17 series amounting to approx. one year of treatment compared to patients who are not treated with trastuzumab.

ELIGIBILITY:
General inclusion criteria:

* Female
* Age > 18 years
* Histologically confirmed breast cancer
* No prior neoadjuvant treatment
* Estrogen receptor positive (>1%)
* Presence of cold activated brown fat as evidenced by a change in Δtemp. of >1°C (post cooling - precooling temperature).

HER2 positive group: HER2-positive (HER2+) and Estrogen receptor-positive (ER+) breast cancer patients (N = 15):

* HER2 positive breast cancer as defined by ASCO/CAP criteria
* Scheduled to receive adjuvant chemotherapy, a total of 17 series of trastuzumab and endocrine treatment

Control group: HER2-negative breast cancer patients (HER2-) and Estrogen receptor-positive (ER+) breast cancer patients (N = 15):

* HER2 negative breast cancer as defined by ASCO/CAP criteria
* Scheduled to receive adjuvant chemotherapy and endocrine treatment

Exclusion Criteria:

* Any other cancer (excluding carcinoma in situ and radically operated localised squamous skin cancer) with clinical activity within the last 2 years
* Metastatic breast cancer
* Metabolic diseases such as diabetes (exceptions can be made if the disease is well treated, assessed by the clinically responsible medical doctor (see section 18))
* Regular use of prednisolone - use in relation to chemotherapy only is ok
* Pregnancy
* Untreated or dysregulated hypertension defined as outpatient clinic systolic BP > 155 and diastolic BP > 95
* Clinically significant ventricular or atrial arrhythmia
* Untreated coronary artery disease or angina pectoris
* Symptomatic heart failure (NYHA ≥ 2)
* Known cold urticaria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed breast cancer (HER2+/HER2-/ER+) sheduled for adjuvant treatment at Rigshospitalet, Copenhagen, Denmark
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
BAT activity | One year
  Difference in cold-induced BAT activity between HER2+ breast cancer patients and HER2- breast cancer controls measured with infrared thermography (temperature difference).

SECONDARY OUTCOMES:
Change in weight | One year
  Difference in weight (kilograms) between the HER2+ positive subjects and the HER2 negative controls
Change fat mass | One year
  Difference in fat mass (kilograms) between the HER2+ positive subjects and the HER2 negative controls
Resting energy expenditure | One year
  Difference in resting- and cold induced energy expenditure (calories/day) between the HER2+ positive subjects and the HER2 negative controls, by measuring oxygen consumption (VO2) and carbon dioxide production (VCO2) (Indirect calorimetry).
Cold induced energy expenditure | One year
  Difference in cold induced energy expenditure (calories/day) between the HER2+ positive subjects and the HER2 negative controls, by measuring oxygen consumption (VO2) and carbon dioxide production (VCO2) (Indirect calorimetry).
Glycemic control (OGTT) - Insulin | One year
  Difference in glycemic control between the HER2+ positive subjects and the HER2 negative controls. Examined by an Oral Glucose Tolerance Test measuring insulin (pmol/L)
Glycemic control (OGTT) - Glucose | One year
  Difference in glycemic control between the HER2+ positive subjects and the HER2 negative controls. Examined by an Oral Glucose Tolerance Test measuring glucose (mmol/L).
Glycemic control (OGTT) - C-peptide | One year
  Difference in glycemic control between the HER2+ positive subjects and the HER2 negative controls. Examined by an Oral Glucose Tolerance Test measuring C-peptide (nmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Søren Nielsen, MSc., Ph.D., Principal Investigator — Centre for Physical Activity Research, Rigshospitalet, University of Copenhagen, Denmark
Locations (1):
- Centre for Physical Activity Research (CFAS), Rigshospitalet, University of Copenhagen, Copenhagen, Denmark